CLINICAL TRIAL: NCT01496027
Title: A Comparison of Cerebral Tissue Oxygenation Values in Newborns Measured Simultaneously Using Laser and LED NIRS Oximeters
Brief Title: Cerebral Tissue Oxygenation Values in Newborns Measured Using Laser and LED NIRS Oximeters
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Tomasz Szczapa, M.D., Poznan University of Medical Sciences
Other Study IDs: 04515
Record Dates: First submitted 2011-12-10; First posted 2011-12-21 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Cerebral Oxygenation
Keywords: cerebral oxygenation; NIRS; tissue oximeters; near infrared spectroscopy; newborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- term newborns
- Preterm Newborns (32-37 GA)

SUMMARY:
The aim of the study is to compare the values of cerebral tissue oxygenation measured simultaneously using laser light (FORE-SIGHT) and LED (INVOS) cerebral oximeters.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable
* Spontaneously breathing newborns

Exclusion Criteria:

* Congenital heart defects or anomalies of central nervous system
* Prematurity below 32 GA
* Respiratory distress

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Clinically stable, spontaneously breathing newborns will be included in the study. Enrolled patients will be divided into two groups: 15 term (≥37 weeks GA) and 15 preterm (32-37 weeks GA) newborns. NIRS measurements will be performed on the 1st and 3rd day of life.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Comparison of variability and repeatability of the recorded cerebral tissue oxygenation signals between two groups of patients (clinical stable preterm and term newborns) | 6 hours
  There are two FDA-approved near infrared cerebral oximeters:
  1. FORE-SIGHT- which uses laser light
  2. INVOS 5100- which uses light emmiting diode.
  Measurements in adult patients have showed that FORE-SIGHT provides more stable signal. Purpose of our study is to compare these two devices in newborn patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Katedra Neonatologii, Poznan, Greater Poland Voivodeship, Poland

REFERENCES:
- [Background] MacLeod D; Ikeda K; Vacchiano C Simultaneous Comparison of FORE-SIGHT and INVOS Cerebral Oximeters to Jugular Bulb and Arterial Co-Oximetry Measurements in Healthy Volunteers ANESTH ANALG 2009; 108(SCA Suppl);1-104